CLINICAL TRIAL: NCT07185074
Title: Effect of Lidocaine Aerosol Combined With Low-dose Cisatracurium vs. Conventional-dose Cisatracurium on Intubation Condition in Patients Undergoing ERCP: a Randomized Clinical Trial
Brief Title: Effect of Lidocaine Aerosol Plus Low-dose Cisatracurium vs Conventional-dose Cisatracurium on Intubation Conditions in ERCP - A Randomized Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangang Song (Other)
Responsible Party: Sponsor-Investigator, Jiangang Song, Study Director, ShuGuang Hospital
Organization: ShuGuang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERCP20240808
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Intubation, Intratracheal
Keywords: cisatracurium; Topical Anesthesia / Aerosol; Lidocaine; ERCP; Noninferiority Trial; Hepatic Dysfunction
MeSH Terms: conditions — Liver Diseases | interventions — cisatracurium

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to allocation. Care providers and investigators who prepare drugs and perform intubation are not blinded. Intubation conditions (Cooper score) are rated by the intubating anesthesiologist (unblinded). Objective secondary outcomes (e.g., intubation time, first-pass success, hemodynamic thresholds) are included to mitigate assessment bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose cisatracurium plus topical lidocaine aerosol (Experimental): Induction with propofol 2.5 mg/kg IV, sufentanil 5 mcg IV, remifentanil 2 mcg/kg IV, and cisatracurium 0.05 mg/kg IV. After approximately 2 minutes, the glottis is exposed with a video laryngoscope and 2.4% lidocaine aerosol is sprayed three times onto the vocal cords. Intubation is performed approximately 3 minutes after induction.
  Interventions: Drug: Cisatracurium 0.05 mg/kg IV; Drug: Lidocaine aerosol 2.4% topical
- Conventional-dose cisatracurium (Active Comparator): Same induction without topical lidocaine; cisatracurium 0.15 mg/kg IV. Intubation approximately 3 minutes after induction using a video laryngoscope.
  Interventions: Drug: Cisatracurium 0.15 mg/kg IV

INTERVENTIONS:
Drug: Cisatracurium 0.05 mg/kg IV — Single bolus at induction; used in the experimental arm. Approximate potency reference: 0.05 mg/kg is about 1 x ED95.
  Arms: Low-dose cisatracurium plus topical lidocaine aerosol
Drug: Cisatracurium 0.15 mg/kg IV — Single bolus at induction; used in the active comparator arm. Approximate potency reference: 0.15 mg/kg is about 3 x ED95.
  Arms: Conventional-dose cisatracurium
Drug: Lidocaine aerosol 2.4% topical — Three sprays to the glottic area immediately before intubation; used only in the experimental arm.
  Arms: Low-dose cisatracurium plus topical lidocaine aerosol

SUMMARY:
This clinical study investigates the effects of lidocaine aerosol as an adjunct to low-dose cisatracurium for endotracheal intubation during ERCP (Endoscopic Retrograde Cholangiopancreatography) procedures. The aim is to assess whether lidocaine aerosol can improve the clinical conditions of intubation to a level comparable to the standard dose of cisatracurium, while reducing the amount of muscle relaxant required. The study also seeks to evaluate the impact of this approach on intubation success, extubation time, and recovery time in the operating room, ultimately improving the efficiency of the operating room. Participants will be randomly assigned to either the low-dose cisatracurium group with lidocaine aerosol or the standard-dose cisatracurium group. The primary outcome is the incidence of clinically acceptable intubation conditions, defined by the Cooper's grading system.

DETAILED DESCRIPTION:
Retrospective registration note. Enrollment began on January 17, 2025, was temporarily paused due to investigator training, and is being reactivated at the time of registration. No changes were made to the prespecified primary outcome or analysis plan. This single-center, randomized (1:1), single-blind trial in adult ERCP patients compares low-dose cisatracurium (≈0.05 mg/kg) plus topical lidocaine aerosol versus conventional-dose cisatracurium (≈0.15 mg/kg). Intubation is performed with a video laryngoscope ~3 min after induction. Primary outcome: clinically acceptable intubation conditions (Cooper score ≥6) at the intubation attempt; key secondary outcomes include intubation time, first-pass success, procedure/OR times, extubation time, and safety through 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled ERCP under general anesthesia requiring endotracheal intubation.
* Hepatic dysfunction: Child-Pugh class B or C.
* Age 18-70 years.
* ASA physical status I-III.

Exclusion Criteria:

* Severe cardiovascular, cerebrovascular, or respiratory disease judged by investigators to increase risk.
* Predicted difficult airway (e.g., Mallampati IV, mouth opening <3 cm, limited neck extension).
* Suspected gastrointestinal obstruction on preoperative assessment.
* Cervical spine disease with limited neck mobility.
* Child-Pugh class C with hepatic encephalopathy.
* Neuromuscular disease.
* Recurrent laryngeal nerve injury or vocal cord dysfunction.
* Pregnancy or breastfeeding.
* Known allergy/hypersensitivity to any study anesthetic (e.g., cisatracurium, lidocaine, propofol, remifentanil, or sufentanil).
* Refusal to participate in the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically acceptable intubation conditions (Cooper score ≥6) | At the intubation attempt following induction (~3 minutes after induction)
  Intubation conditions are graded with the Cooper scale (jaw relaxation, vocal cords, response to intubation; each 0-3). Scores ≥6 are counted as clinically acceptable. Assessed by the intubating anesthesiologist (unblinded).

SECONDARY OUTCOMES:
Intubation time (seconds) | From laryngoscope blade passing the incisors to capnography confirmation of tracheal intubation
  Time in seconds measured with a stopwatch.
First-pass success rate | At the intubation attempt following induction
  Proportion of participants with successful tracheal intubation on the first attempt without rescue cisatracurium.
Procedure duration (minutes) | From endoscope insertion to scope removal (skin-to-skin for ERCP)
  Duration recorded from OR system or anesthesia record.
Extubation time (seconds) | From turning off volatile anesthetic to tracheal tube removal
  Time in seconds measured with a stopwatch.
Operating-room time after ERCP | From scope removal to leaving the operating room
  Duration in minutes.
Severe hemodynamic reaction within 10 minutes after induction | From induction to 10 minutes after induction
  Incidence of HR <45 bpm or >110 bpm or SBP <80 mmHg or >160 mmHg, or need for vasoactive rescue per protocol.
Oxygen desaturation events | From induction to PACU discharge
  Number of participants with SpO₂ ≤92% lasting ≥10 seconds or requiring assisted ventilation.
Airway complications related to intubation | From tracheal intubation to 24 hours after the end of anesthesia.
  Visible blood on laryngoscope, laryngospasm/stridor, re-intubation, or need for airway interventions.
Postoperative nausea and vomiting (PONV) within 24 hours | 0-24 hours after surgery
  Presence of nausea and/or vomiting requiring antiemetic therapy.
Sore throat or hoarseness within 24 hours | 0-24 hours after surgery
  Patient-reported symptoms assessed via standardized questionnaire (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Song, MD, Study Director — Department of Anesthesiology, Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, China
Locations (1):
- Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No